CLINICAL TRIAL: NCT02254915
Title: A Multi-Centre, Randomised, Open-Label Active-Controlled Study Comparing Safety and Efficacy of Synergo Radiofrequency (RF)-Induced Hyperthermia-Chemotherapy With Mitomycin C (RITE) Versus Bacillus Calmette-Guérin (BCG) as First-Line Treatment of Non-Muscle Invasive Papillary Bladder Cancer (NMIBC)
Brief Title: SHTC - EUROPE-1 Synergo Hyperthermia-Chemotherapy by European Urologists' Research Operation Preserving Evolution Study I
Acronym: SHTC-EUROPE-1
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Shortages of the active comparator drug (BCG) on the market worldwide and a growing uncertainty as to its future supply.
Sponsor: Medical Enterprises Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-002-00
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms; Neoplasms by Site; Urinary Bladder Diseases; Urologic Diseases
Keywords: Synergo; RITE; SHTC; Non Muscle Invasive Bladder Cancer; NMIBC; Superficial Bladder Cancer; Urothelial Cell Cancer; Transitional Cell Cancer; Mitomycin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms; Neoplasms by Site; Urinary Bladder Diseases; Urologic Diseases; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synergo + MMC (Experimental): Synergo radiofrequency (RF)-Induced hyperthermia-chemotherapy (SHTC) with mitomycin C (RITE) intravesical therapy as first-line adjuvant treatment for intermediate and high-risk NMIBC,
  Interventions: Device: Synergo + MMC
- Bacillus Calmette-Guérin (Active Comparator): Intravesical BCG therapy as first-line adjuvant treatment for intermediate and high-risk NMIBC,
  Interventions: Drug: Bacillus Calmette-Guérin

INTERVENTIONS:
Device: Synergo + MMC — Synergo radiofrequency (RF)-Induced hyperthermia-chemotherapy with mitomycin C (RITE). Intravesical instillation of MMC utilizing the Synergo system.
  Other Names: RITE; SHTC
  Arms: Synergo + MMC
Drug: Bacillus Calmette-Guérin — Intravesical instillation of BCG.
  Other Names: BCG
  Arms: Bacillus Calmette-Guérin

SUMMARY:
A multi-institutional, prospective, randomised, open-label, superiority, comparative, active-controlled, phase 3 study. The study will compare Synergo RF-induced hyperthermia-chemotherapy (SHTC) plus mitomycin C (MMC) to standard treatment of bacillus Calmette-Guérin (BCG) therapy as first-line adjuvant treatment for intermediate and high-risk NMIBC, and will evaluate recurrence and progression rate over two years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary intermediate or high-risk papillary NMIBC according to the EAU Guidelines and intermediate and high-risk recurrences that have not received BCG within the previous 2 years or chemotherapy treatment (apart from one early instillation) within the previous year.
2. All clinical, intra-operative and pathological items for the EAU risk stratification must be documented including a bladder map.
3. Patients must have undergone a re-resection (second TURB in accordance with the EAU Guidelines) (i) if the initial TURB was incomplete (ii) if there was no muscle in the specimen after the initial TURB (except in TaG1/LG tumours) (iii) in all T1 and all G3/HG tumours TURB of T1 sites must include muscle. Re-resection must be negative in patients diagnosed with T1 and/or G3/HG and/or multiple tumours in the initial TURB.
4. No UC in the upper tract, kidney and ureters. This should be confirmed by CT-IVU or IVU performed at time of initial diagnosis in selected cases as recommended in latest EAU guidelines published prior to screening.
5. No UC in the urethra, excluded by visual inspection during cystoscopy and, in addition, in patients with (i) tumour of trigone (ii) tumour of bladder neck (iii) abnormal prostatic urethra UC must be excluded by biopsy of the prostatic urethra in all male patients or, in female patients, from the portion of the urethra adjacent to the bladder neck, before study recruitment.
6. All patients must have urine cytology dated within the screening period prior to randomisation.
7. Age ≥ 18 yrs
8. Normal kidneys and ureters.
9. Pre-treatment haematology and biochemistry values within acceptable limits:

   (i) haemoglobin ≥ 10 g/dl (g/100 ml) (ii) platelets ≥ 150 x 109/L (103/mm3) (iii) WBC ≥ 3.0 x 109/L (103/mm3) (iv) ANC ≥ 1.5 x 109/L (103/mm3, absolute neutrophil count) (v) Serum creatinine, SGOT, SGPT, Alkaline phosphatase: < 1.5 x UNL (upper normal limit)
10. Negative pregnancy test for women of child-bearing potential
11. A life expectancy at least of the duration of the trial.
12. Unfit or unwilling to have a full or partial cystectomy.
13. Signed informed consent.

Exclusion Criteria:

1. UC involving the prostatic urethra
2. Non-UC tumour of the urinary tract
3. Upper tract and intramural tumours (e.g. in Ostium).
4. History of stage > T1 UC.
5. CIS (suspected or present).
6. Known or suspected reduced bladder capacity. Patients will have a US estimation of maximum bladder capacity or void spontaneously the maximum they can retain in their bladder, and this will be used to determine urine volume. A minimum volume of 250 ml is required.
7. Bleeding disorder
8. Macrohaematuria of ≥ 250 RBC's/uL or equivalent (e.g. > "+++" erythrocytes in a dipstick analysis).
9. Pregnant or lactating women.
10. Women of childbearing potential unwilling or unable to use adequate contraception if sexually active.
11. More than a maintenance dose of oral corticosteroids (maintenance dose defined as the same dose regimen over the past 6 months for a condition requiring continual corticosteroid treatment) or patients with an immuno-compromised state for any reason.
12. More than low-dose Methotrexate (>17.5 mg once a week).
13. Other malignancy within the past five years, except: non-melanomatous skin cancer cured by excision, adequately treated carcinoma in situ of the cervix or ductal CIS (DCIS)/lobular CIS (LCIS) of the breast or stable prostate cancer (under active surveillance or hormone control) with a life expectancy of more than 5 years.
14. Any known allergy or adverse event that would prevent them from receiving a treatment that they may be randomised to within the trial.
15. Known untreated strictural disease or bladder neck contracture or any other condition that may prevent catheterisation with 21F catheter. Patients may undergo dilation or urethral incision before entering the study.
16. Bladder diverticula with cumulative diameter > 1cm
17. UTI at any time within 6 months preceding randomisation.
18. Significant urinary incontinence (spontaneous, requiring use of pads)
19. History of pelvic irradiation
20. Patients with implanted electronic devices (such as cardiac pacemakers) unless they receive permission from their treating physician (e.g., cardiologist) and are monitored by a treating physician during the treatment session.
21. Participation in another study which includes treatment that is liable to have an effect on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
RFS time | 2 years
  The recurrence-free survival time in patients with NMIBC following treatment with SHTC (investigational arm) compared to BCG (controlled arm).

SECONDARY OUTCOMES:
Progression-free survival time | 2 years
Recurrence free survival time by risk group | 2 years
Organ preservation rate | 2 years
Overall survival time | 2 years
Disease-specific survival time | 2 years
Adverse events | 2 years
  Safety (rate of adverse events), as well as tolerability of SHTC compared to BCG in terms of the frequency, severity and nature of adverse events and the treatment received.
Treatment discontinuation | 2 years
  Proportion of treatment discontinuation of SHTC compared to BCG

CONTACTS AND LOCATIONS:
Overall Officials: Igal Ruvinsky, PhD, Study Director — Medical Enterprises Europe B.V.; Gerson Luedecke, Dr. med., Principal Investigator — Universitätsklinikum Gießen und Marburg